CLINICAL TRIAL: NCT03889496
Title: Quantitative GLP-1 Receptor Imaging Correlated to ex Vivo Distribution of In-111-exendin
Acronym: GLP1-ex-vivo
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Because of the COVID-19 pandemic, funding for the trial was terminated and attempts to find alternative sources of funding were to no avail.
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NL47132.091.14
Record Dates: First submitted 2019-01-23; First posted 2019-03-26 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2020-10

CONDITIONS: Diabetes Mellitus
Keywords: exendin-4; GLP-1 receptor imaging; SPECT; pancreas; surgery; quantification
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Scheduled for (partial) pancreatectomy or Whipple procedure (Other): I.v. injection with In-111-DTPA-exendin-4 and SPECT/CT scan
  Interventions: Radiation: indium-111-exendin SPECT/CT

INTERVENTIONS:
Radiation: indium-111-exendin SPECT/CT — SPECT/CT imaging after injection with In-111-DTPA-exendin-4

SUMMARY:
The main goal is to study the correlation of pancreatic uptake of In-111-DTPA-exendin-4 (measured by ex vivo counting) with the beta cell mass determined in the pancreatic specimens obtained after surgery.

DETAILED DESCRIPTION:
In order to fully characterize the highly promising tracer In-111-DTPA-exendin-4 in humans, quantitative SPECT imaging will be correlated to the ex vivo tracer distribution in patients undergoing pancreatectomy or a Whipple procedure. In vivo imaging will be combined with post-pancreatectomy (micro)autoradiography, measurement of In-111-DTPA-exendin-4 concentrations in the pancreas using a gamma counter and morphometric determination of the actual beta cell mass. By this means, the relation between tracer uptake and beta cell mass in non-diabetic patients and T2D patients will be established. These highly relevant data will allow the improvement of the interpretation of clinical quantitative SPECT data in subsequent studies in patients with T1D and T2D. In addition, high uptake has been observed in the duodenum/pyloric area in patients in an ongoing study. At this point in time, it remains unclear which cells are responsible for this uptake. It would be of great interest to identify the GLP-1R positive cells in order to better understand the physiological actions of GLP-1 agonists.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for partial or complete pancreatectomy or Whipple procedure at Radboudumc

Exclusion Criteria:

* Resection that provides insufficient amount of tissue
* Previous treatment with synthetic Exendin (Exenatide, Byetta®) or Dipeptidyl- Peptidase IV inhibitors
* Breast feeding
* Pregnancy or the wish to become pregnant within 6 months
* Renal disease
* Liver disease
* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-11-16 (Actual); Primary Completion 2021-06-14 (Actual); Study Completion 2021-06-14 (Actual)

PRIMARY OUTCOMES:
Correlation between the tracer uptake (counts) and beta cell mass (mg) | 4 years
  The primary objective is the correlation between the ex vivo In-111-exendin tracer accumulation in the pancreas (counts) of patients undergoing pancreatectomy or Whipple procedure, and the beta cell mass (mg) in non- diabetic patients and patients with diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Gotthardt, Prof. Dr., Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud university medical center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jansen TJP, Tokgoz S, Buitinga M, van Lith SAM, Joosten L, Frielink C, Smeets EMM, Stommel MWJ, van der Kolk MB, de Galan BE, Brom M, Boss M, Gotthardt M. Validation of radiolabelled exendin for beta cell imaging by ex vivo autoradiography and immunohistochemistry of human pancreas. EJNMMI Res. 2024 Oct 15;14(1):96. doi: 10.1186/s13550-024-01159-6. PMID 39405026